CLINICAL TRIAL: NCT06168799
Title: Double-Blind, Randomized, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Ilofotase Alfa in Patients at Risk for Renal Damage Following Open Heart Surgery
Brief Title: Ilofotase Alfa for Prevention of Renal Damage After Cardiac Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AM-Pharma (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AP-recAP-CSA-RD-02-01; WHO Universal Trial Number (Registry Identifier: U1111-1295-0827); EU Clinical Trial Number (Registry Identifier: 2023-505859-45)
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Open Heart Surgery
Keywords: Renal; Kidney; Cardiac; CPB; CABG

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ilofotase alfa (Experimental)
  Interventions: Drug: Ilofotase alfa
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ilofotase alfa — After dilution of the concentrate, the investigational medicinal product will be administered by intravenous infusion for 1 hour at the same day before and after the surgery (Day 1)
  Arms: Ilofotase alfa
Drug: Placebo — After dilution of the concentrate, the investigational medicinal product will be administered by intravenous infusion for 1 hour at the same day before and after the surgery (Day 1)
  Arms: Placebo

SUMMARY:
The aim of this clinical trial is to evaluate the efficacy and safety of two intravenous administrations of ilofotase alfa in patients at risk for renal damage following open heart surgery.

DETAILED DESCRIPTION:
This is a Phase 2, multi-center, randomized, double-blind, placebo-controlled, 2-arm parallel group design trial in patients at risk for renal damage following open heart surgery. After screening and baseline assessments, eligible patients will be randomized 1:1 to either 2 doses of 128 mg ilofotase alfa, or 2 doses of placebo control. Randomization will be stratified by baseline eGFR and type of surgery. The patient will be treated with the investigational product (ilofotase alfa or placebo) at the same day before and after the surgery (Day 1). Follow-up clinic visits will be performed daily up to Day 5 for efficacy, safety, and pharmocokinetics assessments. A safety follow-up can be performed by telephone at Day 28. At Day 61, an end of trial visit will be done at site for efficacy, safety, and anti-drug antibodies assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Planned for one of the following types of open chest cardiovascular surgery with the use of cardiopulmonary bypass pump (CPB):

   1. 1. combined valve and CABG surgery; 2. aortic valve plus aortic root and/or ascending aorta (excluding aortic arch)
   2. CABG with 3 or more distal anastomoses
3. Screening eGFR ≥25 mL/min/1.73m2 and ≤65 mL/min/1.73m2
4. Female patients of childbearing potential agreeing to use effective contraception within IP treatment and 14 days thereafter

   Post-menopausal females do not require contraception during the trial.
5. Male patients agreeing to refrain from donating sperm, use a male condom when having sexual intercourse and in case their partner is of childbearing potential they must agree to use adequate and effective contraception method (see inclusion criterion 4) within IP treatment and 14 days thereafter

The five most important Exclusion Criteria:

1. Body weight ≤55 kg
2. Known or suspected glomerulonephritis (other than diabetic kidney disease) or other systemic vasculitis
3. Confirmed or treated endocarditis requiring antimicrobial or antiviral treatment within 30 days prior to surgery or other current active infection requiring antimicrobial or antiviral treatment within 14 days prior to surgery
4. Known chronic liver disorder with Child-Pugh C classification
5. Current planned (or scheduled) surgical intervention under conditions of circulatory arrest, including planned deep hypothermic circulatory arrest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 271 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2025-10-05 (Actual); Study Completion 2025-12-03 (Actual)

PRIMARY OUTCOMES:
Assessment of serum creatinine values | From Baseline to Day 5
  Ratio between the highest value postsurgery (post-surgery Day 1 and Days 2, 3, 4, and 5) and the pre-surgery baseline value for serum creatinine

SECONDARY OUTCOMES:
Assessment of major adverse kidney events (MAKE) 60 | Daily post-surgery through Day 5
  Major adverse kidney events (MAKE) 60, defined as died up to and including Day 61, have received or are receiving new renal replacement therapy (RRT) up to and including Day 61, or have a decrease in estimated glomerular filtration rate (eGFR) ≥25% on Day 61 compared to the pre-surgery baseline eGFR reference value
Assessment of adverse event (AE) and serious adverse event (SAE) occurrence | From Day -1 to Day 28

OTHER OUTCOMES:
AUC of AKI | From Day 1 to Day 5
  The area under the curve (AUC) of acute kidney injury (kidney disease improving global outcomes [KDIGO] sCreat), defined as duration (in days) and severity of acute kidney injury (AKI); measured over the first 5 days after surgery
Incidence of KDIGO AKI | From Day 1 to Day 5
  The overall incidence of KDIGO AKI over the first 5 days after surgery
Assessment of surgery-related complications occurrence | From Day 1 to Day 28
  Postoperative surgery-related complications within 28 days of surgery, assessed according to the Society of Thoracic Surgeons (STS) definition
Assessment of length of stay in the intensive care unit | From Baseline to Day 28
  Length of stay in the intensive care unit (ICU) in days after the initial surgery
Investigation of biomarkers of AKI (optional after the end of the trial) | Pre-surgery Baseline, Day 1 post-surgery, Day 2, Day 3, Day 4, Day 5, and Day 61
  Changes in biomarkers of AKI (urine and blood) compared to Baseline: sCreat, cystatin C and potentially further biomarkers of AKI
Serum levels of ilofotase alfa | Day 1 postsurgery, Day 2, Day 3, Day 4, and Day 5
  Population (Pop) PK

CONTACTS AND LOCATIONS:
Overall Officials: Pickkers, Prof, MD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Research site, Munich, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tellez Garcia JM, Steenvoorden T, Bemelman F, Hilhorst M, Tammaro A, Vogt L. Purinoreceptor P2X7 in Extracellular ATP-Mediated Inflammation through the Spectrum of Kidney Diseases and Kidney Transplantation. J Am Soc Nephrol. 2025 Mar 28;36(9):1823-1843. doi: 10.1681/ASN.0000000711. PMID 40152923